CLINICAL TRIAL: NCT06109142
Title: Pilot Study on the Effect of Oxiris Haemofiltration Membrane on Haemodynamic Stabilisation and Clearance of Vasoactive Metabolites
Brief Title: Clearance of Vasoactive Metabolites With Blood Purification
Acronym: VITAL
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230001; 2022-A01439-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-10-02; First posted 2023-10-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Critically Ill Patients
Keywords: Intensive care; Septic shock; Inflammatory mediators; Renin Angiotensin System
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood - Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extracorporeal blood purification is a supportive therapy in the management of patients with sepsis or vasoplegic shock. The pathophysiology of sepsis is based on an inappropriate host response to infection. Certain medical devices with higher adsorption capacity make it possible to limit this inappropriate response and could thus improve the hemodynamics of patients in septic or vasoplegic shock. The preliminary experience of the investigators from clinical data of vasopressor withdrawal in pediatric patients treated with oXiris shows a 50% reduction in the vasopressor score, Vaso Inotropic Score (VIS), for 40% of patients within 24 hours following the start of treatment. Similar results were found in adult patients treated for severe COVID-19 or vasoplegic shock by the other centers participating in the study.

Cytokine purification is an important physiological effect of purification membranes. However, this may not fully explain the rapid hemodynamic improvement of patients treated with an oXiris membrane.

The role of angiotensin metabolites (Ang 1-5, 1-7, 1-9) in the systemic vascular tone of patients has been recently discussed. The administration of angiotensin 2 in vasoplegic shock in adults helps correct hypotension. In the group of patients with increased renin, this treatment was associated with a reduction in mortality. Indeed, increased renin associated with dysfunction of Angiotensin Converting Enzyme (ACE) leads to an accumulation of Angiotensin 1 which degrades to Ang 1-7.

The hypothesis f the investigators is that the concentration of Ang 1 and Ang 1-7 is elevated in cases of vasoplegic shock and that the clearance of these vasodilator peptides by blood purification is associated with clinical improvement.

DETAILED DESCRIPTION:
This is a pilot study, non-interventional research involving the human subjects, category 3, aimed at measuring the clinical and biological the clinical and biological effects of using the oXiris hemofiltration hemofiltration membrane.

As part of the treatment: oXiris membrane hemofiltration with Prismaflex system, Phoxylium or Hémosol B0 dialysis solution, upper or lower dialysis catheter. Anticoagulation with heparin, citrate or none in case of severe haemostasis disorders. Treatment volume of 35 ml/kg/h maximum.

For research purposes: collection of additional blood tubes (2 x 5mL heparinized tube) added to the usual samples, at the following times:

Baseline (before starting treatment), under hemofiltration at 24h +/- 6h of treatment and at 72 hours +/- 12 hours.

These samples will be analyzed by liquid chromatography - mass spectrometry / mass spectrometry (LC-MS/MS) by Attoquant diagnostics®, a laboratory specialized in analyses of the Renin-Angiotensin system. The angiotensins assayed are Angiotensin I, II, III and IV, as well as the intermediate peptides (1-5, 1-7, 1-9, 2-10, 2-7 and 3-7) and regulatory enzymes (renin, angiotensin converting enzyme, angiotensin 2-converting enzyme and neprilysin).

Angiotensin metabolites have a very short half-life. Their depends on enzyme activity and degradation by circulating proteases. Two techniques are used to determine circulating concentration rapid treatment with protease inhibitors or the equilibrium technique.

For the equilibrium technique, samples are incubated again to restore metabolite concentration prior to analysis. The samples at 3 time points (Baseline, H24 and H72) are analyzed using the equilibrium. The H24 sample will also be analyzed with a protease inhibitor pre-treatment.

Patients will be monitored for 3 months (90-day mortality) using data collected collected in the course of care.

Data from medical records and biological analyses will be entered into an eCRF. Data management will be carried out throughout the study, to enable baseline freezing and statistical analysis as early as possible after the end of the last patient's follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to intensive care with vasoplegic shock (hemodynamic support by noradrenaline).
* Adult or child ≥ 6 years and 30kg
* Indication for extrarenal purification for acute, chronic renal failure, oliguric hydrosodic overload, refractory metabolic acidosis or severe hydroelectrolyte disorder
* Clinician's decision to use an oXiris hemofilter with blood purification capability
* For adult patients: no opposition from the patient (or person of trust or close friend if the patient is unable to be informed)
* For minor patients: no opposition of the holders of parental authority

Exclusion Criteria:

* No need for hemofiltration.
* Citrate anticoagulation of the hemofiltration circuit
* Inclusion in a category 1 or 2 interventional study protocol. Patients included in category 3 interventional research will be able to participate in the study after assessment by the physician.
* Patient under judicial protection and adults under guardianship or curatorship.
* Patient with no social security affiliation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population for pediatric resuscitation concerns:
  * Patients in septic shock requiring extra-renal purification, i.e. 10-20 patients/year
  * Perioperative liver transplant patients, 20% of whom require extra-renal purification for multi-visceral failure associated with shock vasoplegic (5-10 patients/year)
  For adult resuscitations:
  * Patients in septic shock requiring extra-renal purification, i.e. 10-20% of these patients (30 patients per center per year for 2 centers)
  * Perioperative patients of major abdominal surgery with multi-organ renal failure requiring extra-renal purification (20 patients per year for a center).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
50% reduction in vasoinotropic score within 24 hours of initiation on oXiris. | Baseline - 24 hours
  Vaso-inotropic score calculated at baseline and H24. (Minimum 0 = better outcome)

SECONDARY OUTCOMES:
Evolution of the vaso-inotropic score within 72 hours of management | Baseline - 3 hours - 6 hours - 12 hours - 24 hours - 48 hours - 72 hours
  Vaso-inotropic score calculated at baseline - 3 hours - 6 hours - 12 hours - 24 hours - 48 hours - 72 hours (Minimum 0 = better outcome)
Quantitative determination of angiotensins (Ang I, II, III, IV, 1-5, 1-7, 1-9, 2-7, 2-10 and 3-7) and regulatory enzymes (renin, angiotensin-converting enzyme, angiotensin-converting enzyme 2 and neprilysin). | Baseline - 24 hours - 72 hours
  Dosage of angiotensins (Ang I, II, III, IV, 1-5, 1-7, 1-9, 2-7, 2-10 and 3-7) and regulatory enzymes (renin, angiotensin-converting enzyme, angiotensin-converting enzyme 2 and neprilysin) by LC/MS
Clearance of endothelial permeability markers (soluble E-selectin, thromboxane A2, endothelium-derived relaxing factor, bradykinin). | Baseline - 24 hours - 72 hours
  Dosage of Clearance of endothelial permeability markers (soluble E-selectin, thromboxane A2, endothelium-derived relaxing factor, bradykinin) by RT-PCR
Markers of sepsis-induced immunosuppression expressed by HLA-DR monocytes in flow cytometry and selected cytokines (IL-1 beta, IL-6, IL-8, IL-10, TNF-alpha). | Baseline - 24 hours - 72 hours
  Identification of Markers of sepsis-induced immunosuppression expressed by HLA-DR monocytes in flow cytometry and selected cytokines (IL-1 beta, IL-6, IL-8, IL-10, TNF-alpha) by flow cytometry
Mortality at 90 days | Baseline - 24 hours - 90 days
  the correlation between concentrations of metabolites of angiotensin and 90-day mortality
haemodynamic response (concentrations of metabolites of angiotensin) at 24 hours of treatment with oXiris. | Baseline - 24 hours - 90 days
  the concentrations of metabolites of angiotensin

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tissieres, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Garches hospital, Garches
  - Bicetre hospital, Le Kremlin-Bicêtre
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No